CLINICAL TRIAL: NCT00647426
Title: A Phase II Study of Sorafenib in Combination With Carboplatin and Docetaxel in the First Line Treatment of Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Phase II Study of Sorafenib + Carboplatin and Docetaxel in First Line Treatment of Stage IIIB/IV NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 12506
Record Dates: First submitted 2008-03-25; First posted 2008-03-31 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Stage IIIB/IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Sorafenib; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib + Docetaxel/Carboplatin (Experimental): 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
  Interventions: Drug: Sorafenib + Docetaxel/Carboplatin

INTERVENTIONS:
Drug: Sorafenib + Docetaxel/Carboplatin — 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
  Other Names: Carboplatin: Paraplatin, CBDCA

SUMMARY:
This is an open-label, single institution, phase II study of Sorafenib in combination with docetaxel and carboplatin in patients with advanced non-small cell lung cancer. Docetaxel and carboplatin will be given on day 1 of every three week cycle. Patients will take Sorafenib twice a day on the 1st day of treatment and continue to take the medication every day until progression of disease, prohibitive toxicity, or patient withdrawal from the study. Chemotherapy courses will repeat every 21 days in the absence of disease progression or unacceptable toxicity for a total of four cycles.

DETAILED DESCRIPTION:
Patients will be monitored after every two cycles (6 weeks) for tumor response, stability, or progression by radiographic imaging studies. The primary goal of this study is to determine the clinical response rate of this regimen in patients with advanced lung cancer. Secondary endpoints include time to progression, overall survival, and toxicity. Blood levels of ERK-phosphorylation, activated caspase 3, cyclin D1, anti -cIAP2, p-Akt, and Mcl1 activity will be measured at the beginning, middle and end of therapy to help identify predictors of drug response and toxicity during the first cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC with clinical or radiological evidence of advanced disease (Stage IIIB/IV)
* Uni-dimensionally measurable disease
* Age => 18 years
* ECOG performance status of 0-1
* Life expectancy > 3 months

Exclusion Criteria:

* Small-cell or mixed histologies including a small cell component
* Prior chemotherapy, biotherapy, radiotherapy to an area of measurable disease
* Patients with peripheral neuropathy grade => 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2011-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Evans, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafinb + Docetoxel+Carboplatin: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
  Sorafenib + Docetaxel/Carboplatin: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
Period: Overall Study
Arm/Group | Sorafinb + Docetoxel+Carboplatin
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorafinb + Docetoxel+Carboplatin
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Stage IIIB/IV NSCLC Response Rate to the Combination Therapy of Sorafenib and Docetaxel/Carboplatin
Description: The response rate from the combination therapy of Sorafenib and Docetaxel/carboplatin for patients with Stage IIIB/IV NSCLC.The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria (see section 9.3.1).Tumor Response: Evaluation of target lesions Complete Response (CR): Disappearance of all target lesions Partial Response (PR): a) At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
  Progressive Disease (PD): a) At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 30 months
Population: Sufficient data was not collected.
Groups:
- Sorefenib +Docetaxel: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
  Sorafenib + Docetaxel/Carboplatin: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
Arm/Group | Sorefenib +Docetaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants the Progression-free Survival (PFS) .
Description: Disease progression is based on RECIST documentation. Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: 30 months
Population: Sufficient data was not collected.
Groups:
- Sorafenib+Docetaxel: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
  Sorafenib + Docetaxel/Carboplatin: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
Arm/Group | Sorafenib+Docetaxel
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Assessment of adverse events related to the combination infusion, These include a Serious Adverse Event (SAE) is an adverse event occurring at any dose that results in any of the following outcomes:
  1. Death
  2. Life-threatening
  3. Persistent or significant disability/incapacity
  4. In patient hospitalization or prolongation of existing hospitalization
  5. Congenital anomaly/birth defect or • blood dyscrasia without inpatient hospitalization
     * convulsions without inpatient hospitalization
     * intensive treatment in an emergency room or at home for allergic bronchospasm without inpatient hospitalization
     * development of drug dependency
     * drug abuse
     * overdose with an associated serious event, or required intervention to prevent impairment/damage
Time Frame: 30 months
Population: Sufficient data was not collected.
Arm/Group | Sorefenib +Docetaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: The Number of Participants With Biomarkers of Sorafenib Activity and Toxicity
Description: Monitored at designated timepoints.All patients will be evaluable for toxicity from the time of their first treatment with SORAFENIB.
Time Frame: 30 months
Population: Sufficient data was not collected.
Arm/Group | Sorafenib+Docetaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: MedDRA
Groups:
- Sorafenib + Docetaxel: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
  Sorafenib + Docetaxel/Carboplatin: 400 mg po BID Sorafenib + 75 mg/m2 IV Docetaxel on day 1 plus AUC 6 on Carboplatin on day 1 of each 21 day cycle
Arm/Group | Sorafenib + Docetaxel
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No